CLINICAL TRIAL: NCT01896557
Title: Possible Drug Interaction Between Clopidogrel and Ranitidin or Omeprazole in Patients With Stable Coronary Heart Disease: a Comparative Study
Brief Title: Ranitidin Versus Omeprazole in Patients Taking Clopidogrel
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: InCor Heart Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0136/11
Record Dates: First submitted 2013-06-19; First posted 2013-07-11 (Estimated); Results first posted 2016-05-23 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2011-10

CONDITIONS: Coronary Artery Disease; Drug Interaction Potentiation
Keywords: clopidogrel; omeprazole; ranitidin; interaction; aggregability
MeSH Terms: conditions — Coronary Artery Disease | interventions — Omeprazole; Ranitidine; Clopidogrel; Purinergic P2Y Receptor Antagonists

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- omeprazole (Experimental): Omeprazole 20 mg (oral route) twice a day will be given to the subjects for one week. This intervention will be compared with ranitidin 150 mg (oral route) twice a day.
  Interventions: Drug: omeprazole; Drug: Clopidogrel
- ranitidine (Experimental): Ranitidine 150 mg (oral route) twice a day will be given to the subjects for one week.
  Interventions: Drug: Ranitidine; Drug: Clopidogrel

INTERVENTIONS:
Drug: omeprazole — Influence of omeprazole on clopidogrel pharmacodynamics will be evaluated.
  Other Names: Peprazol; Losec; PPI
  Arms: omeprazole
Drug: Ranitidine — Influence of ranitidine on clopidogrel pharmacodynamics will be evaluated.
  Other Names: Antak; H2 receptor blocker
  Arms: ranitidine
Drug: Clopidogrel — Clopidogrel added to ASA therapy at the first medical visit, Open label 75 mg once a day will be given to all individuals as part of the protocol (since main outcome of interest is clopidogrel effect. Actual comparison arms are double blind ranitidine and omeprazole
  Other Names: Plavix; ADP receptor blocker

SUMMARY:
Previous reports have shown a possible drug interaction between clopidogrel and proton pump inhibitors (PPI´s), which could result in increased number of adverse cardiovascular events among patients on dual antiplatelet therapy(DAPT). Because of this, ranitidin has been proposed as an alternative drug to PPI´s for prophylaxis of gastrointestinal bleeding in patients who need DAPT. The study´s aim is to test the hypothesis that ranitidin doesn´t have any influence on clopidogrel pharmacodynamic.

DETAILED DESCRIPTION:
Study population: 100 patients with Stable Coronary Artery Disease from Heart Institute

Inclusion Criteria:

* Age > 18 years old
* Coronary artery disease, defined as previous myocardial infarction and/or coronary angioplasty and/or Coronary Artery Bypass Graft (CABG) surgery and/or coronariography showing obstruction of at least 50 % in one of major epicardial vessels
* Treatment with Acetylsalicylic Acid (ASA) 100 mg/day

Exclusion Criteria:

* Use in the last 7 days of oral anticoagulant or any other antiplatelet drug beside ASA
* Previous utilization of PPI or ranitidine in the last 7 days before randomization
* Active bleeding
* Pregnancy or woman of childbearing age without contraceptive method
* Hemoglobin < 10 g/dL or hematocrit < 30 %, hematocrit > 50 %, platelets < 100.000/mm3 or > 500.000/mm3; creatinin clearance < 50 ml/minute
* Percutaneous coronary intervention (PCI) on the last 30 days before randomization (or PCI on the last year when drug-eluted stents are used); CABG surgery on the last 90 days; acute coronary syndrome on the last 60 days
* Active malignant neoplasm
* Active peptic ulcer disease on the last 60 days or upper gastrointestinal bleeding any time in life
* Known allergy to the drugs clopidogrel, ranitidine or omeprazole
* Refuse to participate in the study]

Methodology: The study has a double-blind, double-dummy prospective design. Clopidogrel action is evaluated by platelet function tests: VerifyNow, bioimpedance aggregometry and Platelet Function Analyzer-100 (PFA-100). The patients have measurements of platelet function on three moments: before starting clopidogrel; 1 week after DAPT with clopidogrel (without loading dose) plus ASA; and after 1 week of randomization to ranitidin 150 mg bid or omeprazole 20 mg bid.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Coronary artery disease, defined as previous myocardial infarction and/or coronary angioplasty and/or CABG surgery and/or coronariography showing obstruction of at least 50 % in one of major epicardial vessels
* Treatment with Acetylsalicylic Acid (ASA) 100 mg/day

Exclusion Criteria:

* Use on the last 7 days of any other antiplatelet drug beside ASA or oral anticoagulant
* Previous utilization of PPI or ranitidine in the last 7 days before randomization
* Any active bleeding
* Pregnancy or woman of childbearing age without contraceptive method
* Hemoglobin < 10 g/dL or hematocrit < 30 %, hematocrit > 50 %, platelets < 100.000/mm3 or > 500.000/mm3; creatinin clearance < 50 ml/minute
* Percutaneous coronary intervention (PCI) on the last 30 days before randomization (or PCI on the last year when drug-eluted stents are used); CABG surgery on the last 90 days; acute coronary syndrome on the last 60 days
* Active malignant neoplasm
* Active peptic ulcer disease on the last 60 days or upper gastrointestinal bleeding any time in life
* Known allergy to the drugs clopidogrel, ranitidine or omeprazole
* Refuse to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2011-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: José C Nicolau, Professor, Principal Investigator — Director of Acute Coronary Care Unit

REFERENCES:
- [Derived] Furtado RHM, Giugliano RP, Strunz CMC, Filho CC, Ramires JAF, Filho RK, Neto PAL, Pereira AC, Rocha TR, Freire BT, D'Amico EA, Nicolau JC. Drug Interaction Between Clopidogrel and Ranitidine or Omeprazole in Stable Coronary Artery Disease: A Double-Blind, Double Dummy, Randomized Study. Am J Cardiovasc Drugs. 2016 Aug;16(4):275-284. doi: 10.1007/s40256-016-0172-5. PMID 27289472

RESULTS

PARTICIPANT FLOW:
Groups:
- Ranitidine: Ranitidine 150 mg BID oral route was added to clopidogrel.
Period: Clopidogrel Alone
Arm/Group | Omeprazole | Ranitidine
Started | 44 | 48
Completed | 43 | 48
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Clopidogrel + GI Protector
Arm/Group | Omeprazole | Ranitidine
Started | 43 | 48
Completed | 41 | 44
Not Completed | 2 | 4
Not completed — low adherence | 1 | 1
Not completed — Reading error | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omeprazole | Ranitidine | Total
Number analyzed (Participants) | 44 | 48 | 92
Age, Categorical [Count of Participants; unit: Participants] — Age according to categories (bellow versus more than or equal to 65 years-old)
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 24 | 26 | 50
    >=65 years | 20 | 22 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (10.9) | 62.5 (8.9) | 62.6 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 25
  Male | 33 | 34 | 67

OUTCOME MEASURES:

1. Primary Outcome: Comparing Platelet Function of Patients on Dual Antiplatelet Therapy With ASA + Clopidogrel, Between the Groups Ranitidin and Omeprazole, After One Week of Randomized Treatment
Description: One week after starting double-blind, double-dummy, randomized therapy with ranitidin or omeprazole on patients treated with DAPT, platelet function will be compared with the method VerifyNow, in P2Y12 Reactivity Units.
Time Frame: One week after randomized treatment exposure (omeprazole or ranitidine)
Measure: Mean (Standard Deviation); unit: P2Y12 Reactivity Units
Arm/Group | Omeprazole | Ranitidine
Number analyzed (Participants) | 41 | 44
P2Y12 Reactivity Units | 173.54 (72.28) | 153.61 (70.12)

2. Primary Outcome: Comparing Platelet Function of Patients on Dual Antiplatelet Therapy With ASA + Clopidogrel, Between the Groups Ranitidin and Omeprazole, Using VerifyNow Method.
Description: One week after starting double-blind, double-dummy, randomized therapy with ranitidin or omeprazole on patients treated with DAPT, platelet function will be compared with the method VerifyNow, in percent Inhibition of Platelet Aggregation (IPA) from baseline. IPA was calculated as the percent change in aggregability from baseline, with the formula IPA = (on-treatment aggregability minus baseline aggregability)/baseline aggregability. Since baseline aggregation is always, per definition, equal or more than on-treatment aggregation, there is no possibility that this number might be negative.
Time Frame: One week after drug exposure (omeprazole/ranitidine); 2 weeks after baseline
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Omeprazole | Ranitidine
Number analyzed (Participants) | 41 | 44
Percentage | 17.4 (33.1) | 30.1 (31.3)

3. Other Pre Specified Outcome: Comparison of the Primary Outcome With Bioimpedance Aggregometry
Description: After 1 week of randomization to ranitidin or omeprazole, the platelet function will also be analysed by other method: bioimpedance aggregometry with ADP 10 mcM as reagent
Time Frame: 1 week after drug exposure
Population: Platelet aggregation was measured after one week of randomized treatment therapy
Measure: Mean (Standard Deviation); unit: Ohms
Arm/Group | Omeprazole | Ranitidine
Number analyzed (Participants) | 41 | 44
Ohms | 2 (2.55) | 2.77 (3.84)

4. Other Pre Specified Outcome: Comparing the Main Outcome on Pre-specified Subgroups
Description: The main outcome will be compared on pre-specified subgroups:
  * elderly (age > 65 yrs-old) versus non-elderly
  * male versus female
  * smoking versus non-smoking patients
  * obese (BMI > 30 kg/m2) versus non-obese
  * diabetic versus non-diabetic
  * patients in use or not in use of statins
  * presence or not of genetic polymorphisms on cytochrome 2C19.
Time Frame: 1 week after drug exposure
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Comparison of the Primary Outcome With PFA-100 (Collagen/ADP Cartridge)
Description: After 1 week of randomization to ranitidin or omeprazole, the platelet function will also be analysed by other method: PFA-100(Collagen/ADP cartridge).
Time Frame: 1 week after drug exposure
Population: Platelet aggregation by PFA-100 was measured after one week of randomized treatment therapy
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Omeprazole | Ranitidine
Number analyzed (Participants) | 33 | 36
seconds | 95.1 (46.2) | 97.2 (79)

ADVERSE EVENTS:
Arm/Group | Omeprazole | Ranitidine
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/48
Other Adverse Events (participants affected / at risk) | 1/44 | 0/48
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omeprazole (N=44) | Ranitidine (N=48)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) — Dyspepsia after clopidogrel was introduced without GI protector

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No